CLINICAL TRIAL: NCT03227159
Title: Study for Evaluation of Newly Onset Chest Pain and Rapid Diagnosis of Myocardial Necrosis (stenoCARDIA)
Brief Title: Study for Evaluation of Newly Onset Chest Pain and Rapid Diagnosis of Myocardial Necrosis
Acronym: stenoCARDIA
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 837.075.06
Record Dates: First submitted 2017-07-11; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Troponin; Emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A venous blood sample (10 ml EDTA, 10ml Citrate, 10ml Serum) for storage and further analysis
  * A venous blood sample (10 ml EDTA ) DNA Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a national multi-center, prospective surveillance study in patients with suspected acute coronary syndrome. Eligible patients must present to one of the participating Emergency Departments within 24 hours from the time of symptom onset. Approximately 2000 patients >18 and <85 years of age are planned to be enrolled.

Upon enrollment in the Emergency Department, a venous blood sample will be obtained from each patient for analysis. The patient's diagnostic work-up, treatment and disposition will continue per the standards of the treating institution. Results will be recorded for ECGs, any cardiac biomarkers measured at the site and any follow-up cardiac objective tests performed for evidence of coronary artery disease and/or myocardial damage (exercise treadmill, coronary angiography, cardiac thallium or technetium scintigraphy, etc).

The Principal Investigator at each site will evaluate the results of the diagnostic cardiac tests performed for that patient to determine whether each patient enrolled at their site has a final diagnosis of ACS.

The status of each patient will also be assessed at 1 month and 6 months after enrollment for intercurrent Major Adverse Cardiac Events (MACE), including myocardial infarction, cardiac revascularization and death.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who are able to give consent. This has to be carefully verified in each case, by the doctors leading the study
* Men or women >18 and <85 years of age
* Patients with chest discomfort within last 24h and suspected Acute Coronary Syndrome (STEMI, NSTEMI and unstable angina)
* Patient experiencing at least 30 minutes of chest discomfort or other symptoms consistent with possible ACS; (Note: Patients who have symptoms of shorter duration that resolved due to pharmacologic intervention may be included.)
* Written informed consent

Exclusion Criteria:

* Age <18 or >85 years
* Inpatient in the hospital prior to onset of symptoms.
* Obvious traumatic disease
* Prisoners or other institutionalized or vulnerable individuals
* Major surgery within last 4 weeks
* Patients with cardiogenic shock
* Other significant laboratory abnormalities that the investigator feels may compromise the patient's safety by participation in the study
* Women who are pregnant or breast feeding
* Obvious iv drug abuse
* Refusal to provide written informed consent
* Unavailability of a telephone number and insufficient contact information as well as permanent residence abroad
* Unreliability as a study participant as based on the investigator's prior knowledge of the patient, such as the inability or willingness to participate in or complete the study or the presence of concurrent physical or psychological disorders that may make it impractical for the patient to participate in or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on patients presenting to the ED within 24 hours of the onset of chest pain. Both patients then discharged to home as well as patients subsequently admitted to the hospital are eligible for the study and may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1818 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute coronary syndromes | 30 days
  The primary end-point of the study is the early diagnosis of acute coronary syndromes using a combined analysis of multiple markers compared to single marker analyses (final diagnosis of ACS as reason for hospital admission).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, MD, Principal Investigator — University Heart Center Hamburg

REFERENCES:
- [Result] Keller T, Zeller T, Ojeda F, Tzikas S, Lillpopp L, Sinning C, Wild P, Genth-Zotz S, Warnholtz A, Giannitsis E, Mockel M, Bickel C, Peetz D, Lackner K, Baldus S, Munzel T, Blankenberg S. Serial changes in highly sensitive troponin I assay and early diagnosis of myocardial infarction. JAMA. 2011 Dec 28;306(24):2684-93. doi: 10.1001/jama.2011.1896. PMID 22203537
- [Result] Keller T, Zeller T, Peetz D, Tzikas S, Roth A, Czyz E, Bickel C, Baldus S, Warnholtz A, Frohlich M, Sinning CR, Eleftheriadis MS, Wild PS, Schnabel RB, Lubos E, Jachmann N, Genth-Zotz S, Post F, Nicaud V, Tiret L, Lackner KJ, Munzel TF, Blankenberg S. Sensitive troponin I assay in early diagnosis of acute myocardial infarction. N Engl J Med. 2009 Aug 27;361(9):868-77. doi: 10.1056/NEJMoa0903515. PMID 19710485
- [Derived] Haller PM, Sorensen NA, Hartikainen TS, Gossling A, Lehmacher J, Toprak B, Twerenbold R, Richter J, Banko T, Korschid S, Schmidt J, Keller T, Zeller T, Blankenberg S, Westermann D, Neumann JT. Rising and Falling High-Sensitivity Cardiac Troponin in Diagnostic Algorithms for Patients With Suspected Myocardial Infarction. J Am Heart Assoc. 2023 May 16;12(10):e027166. doi: 10.1161/JAHA.122.027166. Epub 2023 May 9. PMID 37158171
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Haller PM, Neumann JT, Sorensen NA, Hartikainen TS, Gossling A, Lehmacher J, Keller T, Zeller T, Blankenberg S, Westermann D. The association of anaemia and high-sensitivity cardiac troponin and its effect on diagnosing myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2021 Dec 18;10(10):1187-1196. doi: 10.1093/ehjacc/zuab066. PMID 34350455
- [Derived] Haller PM, Boeddinghaus J, Neumann JT, Sorensen NA, Hartikainen TS, Gossling A, Nestelberger T, Twerenbold R, Lehmacher J, Keller T, Zeller T, Blankenberg S, Mueller C, Westermann D. Performance of the ESC 0/1-h and 0/3-h Algorithm for the Rapid Identification of Myocardial Infarction Without ST-Elevation in Patients With Diabetes. Diabetes Care. 2020 Feb;43(2):460-467. doi: 10.2337/dc19-1327. Epub 2019 Dec 16. PMID 31843947
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Sorensen NA, Chapman AR, Shah ASV, Anand A, Boeddinghaus J, Nestelberger T, Badertscher P, Mokhtari A, Pickering JW, Troughton RW, Greenslade J, Parsonage W, Mueller-Hennessen M, Gori T, Jernberg T, Morris N, Liebetrau C, Hamm C, Katus HA, Munzel T, Landmesser U, Salomaa V, Iacoviello L, Ferrario MM, Giampaoli S, Kee F, Thorand B, Peters A, Borchini R, Jorgensen T, Soderberg S, Sans S, Tunstall-Pedoe H, Kuulasmaa K, Renne T, Lackner KJ, Worster A, Body R, Ekelund U, Kavsak PA, Keller T, Lindahl B, Wild P, Giannitsis E, Than M, Cullen LA, Mills NL, Mueller C, Zeller T, Westermann D, Blankenberg S; COMPASS-MI Study Group. Application of High-Sensitivity Troponin in Suspected Myocardial Infarction. N Engl J Med. 2019 Jun 27;380(26):2529-2540. doi: 10.1056/NEJMoa1803377. PMID 31242362
- [Derived] Sorensen NA, Neumann JT, Ojeda F, Schafer S, Magnussen C, Keller T, Lackner KJ, Zeller T, Karakas M, Munzel T, Blankenberg S, Westermann D, Schnabel RB. Relations of Sex to Diagnosis and Outcomes in Acute Coronary Syndrome. J Am Heart Assoc. 2018 Mar 10;7(6):e007297. doi: 10.1161/JAHA.117.007297. PMID 29525782